CLINICAL TRIAL: NCT06936800
Title: Pinaverium Bromide Preventing Post Extracorporeal Shock Wave Lithotripsy Pancreatitis and Painful (PBPEP): a Single-center, Double-blind, Randomized, Placebo-controlled Trial.
Brief Title: Pinaverium Bromide Preventing Post Extracorporeal Shock Wave Lithotripsy Pancreatitis and Painful (PBPEP)
Acronym: PBPEP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Department of Gastroenterology, Qilu hospital of Shandong University, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QLCR20240052
Record Dates: First submitted 2025-03-29; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pancreatitis; Pancreatic Duct Stones
Keywords: chronic pancreatitis; pancreatic duct stones; ESWL; Pinaverium bromide; Post-ESWL pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — pinaverium; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pinaverium Bromide (Experimental): Preoperative, intraoperative, and postoperative oral administration of 100mg tid of povidone bromide in p-ESWL
  Interventions: Drug: Pinaverium bromide
- Placebo (Placebo Comparator): Preoperative, intraoperative, and postoperative oral administration of 100mg tid of placebo in p-ESWL
  Interventions: Drug: Placebo for control group

INTERVENTIONS:
Drug: Pinaverium bromide — Preoperative, intraoperative, and postoperative oral administration of 100mg povidonium bromide in P-ESWL
  Arms: Pinaverium Bromide
Drug: Placebo for control group — Preoperative, intraoperative, and postoperative oral placebo 100mg for P-ESWL
  Arms: Placebo

SUMMARY:
This study aims to evaluate whether perioperative pinaverium bromide (a calcium antagonist) reduces post-ESWL complications (pancreatitis, abdominal pain, infection) in chronic pancreatitis patients with pancreatic duct stones ≥5mm. A single-center, randomized, double-blind, placebo-controlled design will be used, with 288 participants allocated to either pinaverium bromide (100mg tid) or placebo before and after p-ESWL.

DETAILED DESCRIPTION:
1. Background:

   * Chronic pancreatitis (CP) has a global incidence of 9.62/100,000, often complicated by pancreatic duct stones (90% of CP patients).
   * p-ESWL is first-line for stones >5 mm but carries risks: pancreatitis (4.35%), abdominal pain (42.65%), and other complications (6.73% overall).
   * Pinaverium bromide relaxes the sphincter of Oddi, reduce intestinal spasms and may mitigate post-ESWL complications.
2. Objectives:

   * Primary: Reduce post-p-ESWL pancreatitis incidence (per Atlanta 2012 criteria).
   * Secondary: Decrease abdominal pain, other complications (bleeding, perforation, infection), and drug-related adverse events.
3. Methods:

   * Design: Single-center, randomized, double-blind, placebo-controlled.
   * Sample size estimation This study used a comparative method of two sample rates in a superior efficacy clinical trial, with a unilateral test level of α=0.025 and a confidence level of 1- β=0.8. Based on the previous research on complications of lithotripsy conducted by our center, the incidence of abdominal pain in patients after the first P-ESWL surgery was approximately 42.65%. According to literature research results, pinaverium bromide can improve the relaxation of the Oddi's sphincter by 30-40%. Previous studies have shown that pinaverium bromide can control postoperative abdominal pain at around 18.75%. In this study, it is assumed that pinaverium bromide can reduce the incidence of abdominal pain after ESWL by 25%, from 42.65% to 17.65%, with a cut-off value of 10%, Nt：Nc=1：1. Based on Pearson chi square test, the required sample size was calculated to be 137 cases/group, totaling 274 cases.

   Considering a rejection rate of 5%, the final required sample size is calculated to be 144 cases/group, totaling 288 cases.

   • Intervention: Experimental Group Protocol

   Preoperative Preparation:

   Fasting: 12 hours before ESWL. Water restriction: 4 hours before surgery.

   Medication:

   Oral pinaverium bromide tablets (100mg tid) administered:

   One day before surgery On the day of surgery One day post-surgery

   Postoperative Monitoring:

   Maintain fasting for 24 hours post-surgery.

   Blood tests at 6h and 24h to assess:

   Amylase, lipase, CBC, PCT, CRP Document abdominal pain scores. If abdominal pain worsens or recurs, perform imaging (e.g., abdominal CT). Control Group Protocol

   Preoperative Preparation:

   Identical to the experimental group (fasting 12h, water restriction 4h before ESWL).

   Placebo Administration:

   Oral placebo (2 tablets tid) given:

   One day before surgery On the day of surgery One day post-surgery

   Postoperative Monitoring:

   Identical to the experimental group (fasting, blood tests, pain scoring, and imaging if needed).

   Endpoint evaluation:

   Patients will be closely monitored during and after surgery, with a mandatory hospital stay of at least 48 hours. Endpoint events, including ESWL-related complications (acute pancreatitis, stone street, bleeding, infection, perforation, or others), will be recorded.

   Outcomes: Pancreatitis incidence, pain scores, complications, lab markers (amylase, CRP), and imaging.

   Statistical Methods Principle: All data were analyzed based on the intention-to-treat (ITT) principle.

   Continuous variables were compared using Student's t-test or Mann-Whitney U test, as appropriate.

   Categorical variables were analyzed using the chi-square test or Fisher's exact test, depending on data distribution.

   A P-value < 0.05 was considered statistically significant.
4. Eligibility Criteria

Inclusion:

Age 18-85, CP with ≥5mm pancreatic duct stones (head predominance).

Exclusion:

1. Requirement for repeat ESWL during the study period.
2. Acute pancreatitis within 3 days prior to ESWL.
3. Poor cardiopulmonary function with anesthesia intolerance.
4. Severe liver disease (e.g., hepatic failure, liver abscess, cirrhosis, ascites).
5. Anticoagulant therapy within 3 days or coagulopathy.
6. Suspected or confirmed pancreatic tumor.
7. Arteriosclerosis or abdominal aortic aneurysm obstructing shockwave transmission.
8. Pregnancy or lactation.
9. Allergy to pinaverium bromide
10. Chronic pinaverium bromide use with discontinuation <3 days before ESWL
11. Declined study participation

Termination Criteria:

1. Inability to complete the ESWL procedure due to any reason after initiation.
2. Non-compliance with the trial protocol by the patient.
3. Voluntary withdrawal from the study. 5. Study Arms

   * Experimental: Pinaverium bromide (100mg tid) pre-/post-ESWL.
   * Control: Placebo controlled. 6. Primary Outcome Measures
   * Incidence and severity of post-p-ESWL pancreatitis (Atlanta 2012 criteria). 7. Secondary Outcome Measures
   * Abdominal pain (frequency, duration, scores).
   * Other complications (infection, bleeding, stone street).
   * Drug-related adverse events (e.g., diarrhea, rash). 8. Timeframe
   * Enrollment: April 2025-April 2027.
   * Completion: December 2027. 9. Contacts and Locations
   * Principal Investigator: [Yanqing Li]
   * Site: Qilu Hospital of Shandong University, China.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited, age range is 18-85 years old (inclusive);
2. Perform P-ESWL treatment for painful chronic pancreatitis with positive pancreatic duct stones ≥ 5mm, mainly located in the head or body of the pancreas.

Exclusion Criteria:

1. Requiring repeat ESWL during the study period.
2. Acute pancreatitis within 3 days prior to ESWL.
3. Severe cardiac/pulmonary dysfunction precluding anesthesia tolerance.
4. Advanced liver disease (e.g., liver failure, cirrhosis, ascites, abscess).
5. Anticoagulant use within 3 days or coagulopathy.
6. Suspected or confirmed pancreatic malignancy.
7. Arteriosclerosis or aortic aneurysm along shockwave transmission path.
8. Pregnancy or lactation.
9. Known allergy to pinaverium bromide.
10. Chronic pinaverium bromide use with <3-day washout period.
11. Declined participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and grading of pancreatitis after P-ESWL (mild, moderate, and severe) | 24-48 hours after pancreatic ESWL procedure
  The definition of postoperative pancreatitis after P-ESWL is based on the 2012 Atlanta criteria. If at least two of the following three criteria are met, the diagnosis can be made: abdominal pain consistent with pancreatitis; Within 24 hours after surgery, amylase or lipase should be at least 3 times the normal upper limit; Imaging examination shows characteristic features of pancreatitis

SECONDARY OUTCOMES:
Incidence of abdominal painful after P-ESWL | 24-48 hours after pancreatic ESWL procedure
  Using the Adult Abdominal Pain NRS Rating Scale (NRS) to record the post-ESWL painful.

OTHER OUTCOMES:
Incidence of other adverse events of p-ESWL | 24-48 hours after pancreatic ESWL procedure
  Including bleeding, perforation, infection, steinstrasse.
  1. Clinical evidence of bleeding Mild: hemoglobin drop <3 g, no transfusion Moderate: Transfusion of ≤ 4 units, no angiographic intervention, or surgery Severe: Transfusion of≥ 5 units or intervention (angiographic or surgical)
  2. Infection Mild: > 38 °C for 24-48 hours Moderate:Requires > 3 days of hospital treatment Severe: Abscess, septic shock, or intervention (percutaneous drainage or surgery)
  3. Steinstrasse Mild: Severe abdominal pain without other post-ESWL complications Moderate: Combined with other complications, or requires > 3 days of hospital treatment Severe: Combined with other complications; hospitalization for > 10 days, or surgery
  4. Perforation Mild: Possible, or very slight leak of fluid, treatable with fluids and suction for ≤3days Moderate: Any definite perforation treated medically for 4-10 days Severe: Medical treatment for > 10 days or intervention (percutaneous or surgical)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu hospital of Shandong University, Jinan, Wenhuaxi Road, China

IPD SHARING:
Plan to Share IPD: No